CLINICAL TRIAL: NCT01394328
Title: Delirium in Persons With Dementia
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Collaborators: Augusta University (Other); Harvard University (Other); Indiana University (Other)
Responsible Party: Principal Investigator, Donna Fick, Professor of Nursing, Penn State University
Other Study IDs: 1R03AG023216-01A1 (NIH)
Record Dates: First submitted 2011-07-11; First posted 2011-07-14 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Delirium Superimposed on Dementia
Keywords: Delirium; Dementia; Confusion Assessment Method; Elderly
MeSH Terms: conditions — Delirium; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Persons with Dementia: Persons with Dementia are identified by the Modified Blessed Dementia Rating Scale and the IQCODE

SUMMARY:
The aims of this study were to identify risk factors associated with delirium in hospitalized persons with dementia, and to describe immediate and post-hospital (1&3 months) trajectory of cognitive decline and associated outcomes in persons with dementia who develop delirium. It was hypothesized that factors such as CNS-active medications, urinary tract infection, stage of dementia, pain, activity level, and dehydration would be associated with an increased risk of delirium and delirium severity in patients with dementia compared to dementia patients without delirium. It was also hypothesized that persons with DSD will have worse outcomes (longer hospital length of stays, decreased functional status, a steeper negative slope of cognitive decline) than dementia patients without delirium. Lastly, it was hypothesized that higher delirium severity would be associated with poorer outcomes in persons with dementia. The long-term objectives were to use the results from this study to design and test an intervention strategy to improve early recognition, management, prevention, and outcomes in persons with DSD.

DETAILED DESCRIPTION:
It is well known that persons with dementia are at increased risk of developing delirium or acute confusional state. Further, current evidence suggests that delirium may worsen the prognosis of dementia, may alter the clinical course and trajectory of cognitive decline, and may be associated with substantially worse long-term outcomes. This study was a prospective cohort study design involving 165 hospitalized subjects with dementia who were 65 and older and included a three month follow up period. Aims for the study included: 1) to identify risk factors for DSD, and 2) to describe post-hospital outcomes and the trajectory of cognitive decline for DSD, which will justify the development of appropriate preventative and management strategies for delirium in patients with dementia. Delirium was assessed daily from admission to discharge and then at one and three month follow-ups. The potential risk factors being examined were 1) polypharmacy (central nervous system-active medications, number of medications, new medications added), 2) physical stressors (urinary tract infection, pain, dehydration), and 3) environmental stressors (bedrest, restraints, room changes). Outcomes were assessed by research study staff blinded to the study aims.

ELIGIBILITY:
Inclusion Criteria:

* Persons with dementia were included if they: a) were on one of the selected medical-surgical units and age 65 years or older; b) spoke English; c) were hospitalized less than 24 hours; and d) met the criteria for dementia. This study included minorities and women.

Exclusion Criteria:

* Persons with dementia were excluded if they: a) had any significant neurological or neurosurgical disease associated with cognitive impairment other than dementia (due to confounding with dementia or DSD), such as parkinson's disease, Huntington's disease, normal pressure hydrocephalus, seizure disorder, subdural hematoma, head trauma or any other known structural brain abnormalities; b) were nonverbal and unable to communicate due to sever dementia (MMSE=0), aphasia, intubation, or terminal illness (since interviews were required for the study); or c) had no family or caregivers to interview (since proxy interviews were required for the study). This study did not exclude persons with pre-existing delirium. In addition, subjects were not excluded on the basis of race or gender.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 165 hospitalized older adults at Mount Nittany Medical Center, age 65 and older with Dementia.
Sampling Method: Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2006-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change in Delirium status during hospital stay | Participants will be assessed daily until discharge (duration of hospitalization), which is expected to be about 5 days
  Confusion Assessment Method (CAM)and Delirium Rating Scale (DRS) were used to measure delirium.
Change in Delirium status at 1 month after discharge | Participants will be assessed 1 month after date of hospital discharge
  Confusion Assessment Method (CAM)and Delirium Rating Scale (DRS) were used to measure delirium.
Change in Delirium status at 3 months after discharge | Participants will be assessed 3 months after date of hospital discharge
  Confusion Assessment Method (CAM)and Delirium Rating Scale (DRS) were used to measure delirium.

SECONDARY OUTCOMES:
Hospitalization Length of Stay | Duration of hospitalization, expected to be about 5 days
Change in Functional Status during hospital stay | Daily until discharge, expected to be about 5 days
  Measured using the KATZ ADL Scale and Lawton Index of Daily Living
Change in Functional Status at 1 month after discharge | Participant will be assessed 1 month after date of hospital discharge
  Measured using the KATZ ADL Scale and Lawton Index of Daily Living
Change in Functional Status at 3 months after discharge | Participant will be assessed 3 months after date of hospital discharge
  Measured using the KATZ ADL Scale and Lawton Index of Daily Living
Change in Cognitive Decline during hospital stay | Daily until discharge, expected to be about 5 days
  MMSE and Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) used to measure cognition
Change in Cognitive Decline at 1 month after discharge | Participant will be assessed 1 month after date of hospital discharge
  MMSE and Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) used to measure cognition
Change in Cognitive Decline at 3 months after discharge | Participant will be assessed 3 months after date of hospital discharge
  MMSE and Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) used to measure cognition

CONTACTS AND LOCATIONS:
Overall Officials: Donna Fick, PhD, Principal Investigator — Penn State University
Locations (1):
- Mount Nittany Medical Center, State College, Pennsylvania, United States